CLINICAL TRIAL: NCT02825641
Title: Premature Rupture of Membranes at Term With an Unfavorable Cervix (Bishop Score<6): Comparison of Oxytocin, Dinoprostone Induction and Expectant Management
Brief Title: Premature Rupture of Membranes With a Bishop Score<6: Comparison of Medical Induction/Expectant Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0213-15-RMB
Record Dates: First submitted 2016-06-06; First posted 2016-07-07 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Medical Induction of Labor Affecting Newborn
MeSH Terms: interventions — Oxytocin; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Expectant Management-Dinoprostone (Active Comparator): Women with premature rupture of membranes who are not in active labor and have an unfavorable cervix (Bishop score<6).
  Labor induction will be initiated with Dinoprostone after 24 hours of waiting depending on obstetric history and cervical conditions.
  Interventions: Drug: Dinoprostone
- Expectant Management-Oxytocin (Active Comparator): Women with premature rupture of membranes who are not in active labor and have an unfavorable cervix (Bishop score<6).
  Labor induction will be initiated with oxytocin after 24 hours of waiting depending on obstetric history and cervical conditions.
  Interventions: Drug: Oxytocin
- Active Management-Dinoprostone (Experimental): Women with premature rupture of membranes who are not in active labor and have an unfavorable cervix (Bishop score<6).
  Labor induction will be initiated with Dinoprostone on presentation depending on obstetric history and cervical conditions.
  Interventions: Drug: Dinoprostone
- Active Management-Oxytocin (Experimental): Women with premature rupture of membranes who are not in active labor and have an unfavorable cervix (Bishop score<6).
  Labor induction will be initiated with oxytocin on presentation depending on obstetric history and cervical conditions.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Labor induction and cervical ripening by oxytocin in women with premature rupture of membranes in 2 types of women:
  1. Induction of labor on presentation at the delivery room.
  2. Induction of labor after 24 hours of rupture of membranes.
  Other Names: Pitocin
  Arms: Active Management-Oxytocin; Expectant Management-Oxytocin
Drug: Dinoprostone — Labor induction and cervical ripening by dinoprostone in women with premature rupture of membranes in 2 types of women:
  1. Induction of labor on presentation at the delivery room.
  2. Induction of labor after 24 hours of rupture of membranes.
  Other Names: Cervidil
  Arms: Active Management-Dinoprostone; Expectant Management-Dinoprostone

SUMMARY:
The study is intended to compare expectant management and on presentation labor induction in women with premature rupture of membranes.

The means of labor induction and cervical ripening are either oxytocin or dinoprostone.

Expectant management in this obstetrical state means waiting 24 hours from the onset of rupture of membranes and then commencing labor induction with either oxytocin or dinoprostone depending on the patient's obstetrical history and cervical condition.

The investigators' hypothesis is that active management will lead to a higher rate of vaginal deliveries, a shorter interval between the time of rupture of membranes and the time of delivery, a lower rate of cesarean sections and a better obstetric result for the mother and the fetus/newborn.

DETAILED DESCRIPTION:
In the setting of premature rupture of membranes in term pregnancies, it is customary in women who are not in active labor to wait for 24 hours before attempting to induce labor. The means of labor induction used at our medical center are either intravenous oxytocin or per-vaginal dinoprostone, depending on patient's obstetric history and cervical conditions.

The investigators hypothesize that commencing induction of labor at presentation in these women by either means of induction will lead to higher rates of vaginal delivery, shorter intervals between the time of onset of rupture of membranes and the time of delivery and lower rates of cesarean sections.

The participants in the study, upon signing informed consents, will be randomized to 4 groups-2 groups of expectant management in which labor induction will be commenced after 24 hours with either oxytocin or dinoprostone and 2 groups of active management in which labor induction will be commenced at presentation with either oxytocin or dinoprostone.

The participants will be followed from the time of presentation with rupture of membranes at the delivery room and until the time of delivery.

Further obstetric, clinical and demographic information will be acquired from the patient's electronic medical file for analysis accuracy and sub-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancies >37 weeks of gestation.
* Certain rupture of membranes.
* Bishop score < 6.
* Singleton pregnancies.
* Vertex presentation.
* No obstetric or clinical contraindications for labor induction.
* Reactive non stress test on presentation.

Exclusion Criteria:

* Previous cesarean section.
* Previous uterine surgeries (Myomectomy etc.).
* Placenta Previa.
* Multiple gestation pregnancies.
* Pregnancies with history of fetal reduction or Intrapartum uterine fetal demise.
* Known fetal defects/Chromosomal abnormalities.
* Active genital Herpes.
* HIV carrier.
* Contractions that are less than 10 minutes apart.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 458 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery rate | Up to 7 days from the time of presentation with rupture of membranes
  The percentage of participants that achieved vaginal delivery

SECONDARY OUTCOMES:
Interval to delivery | Up to 7 days from the time of presentation with rupture of membranes
  Interval from the time of onset of premature rupture of membranes and the time of delivery (In minutes)
Caesarian delivery rate | Up to 7 days from the time of presentation with rupture of membranes
  The percentage of participants that required caesarian delivery

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weissman, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No